CLINICAL TRIAL: NCT00047918
Title: Investigation of Hematologic Parameters in Mastocytosis and Idiopathic Anaphylaxis
Brief Title: Blood Factors in Mastocytosis and Unexplained Anaphylaxis and Flushing
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030010; 03-I-0010
Record Dates: First submitted 2002-10-22; First posted 2002-10-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-08

CONDITIONS: Mastocytosis; Anaphylaxis
Keywords: Mast Cells; Bone Marrow; Flushing; Mutations; Mastocytosis; Anaphylaxis
MeSH Terms: conditions — Mastocytosis; Anaphylaxis; Flushing

SUMMARY:
This study will 1) identify characteristics of bone marrow mast cells in patients with unexplained anaphylaxis and flushing or with mastocytosis and 2) determine whether mastocytosis might be the underlying cause of unexplained anaphylaxis in some patients with this condition. Anaphylaxis is a hypersensitivity reaction in which patients may have flushing, hives, stuffy nose, red itchy eyes, difficulty breathing, swelling of the tongue, throat, palms and soles, abdominal cramping, lightheadedness, decreased blood pressure, and loss of consciousness. Although allergens are a common cause of anaphylactic episodes, no cause can be identified in up to 50 percent of patients who have recurrent events. Mastocytosis is a disease of excessive mast cells in tissues such as skin and bone marrow. These cells can release chemicals that result in itching, blisters, flushing, bone pain, and abdominal pain.

Patients 18 years of age and older who have episodes of anaphylaxis or flushing with no apparent cause or who have mastocytosis may be eligible for this study. Participants will have a medical history and physical examination; blood tests to identify genetic changes that are important in the growth, development, and functioning of human mast cells; and bone marrow aspiration and biopsy. For the bone marrow procedure, the skin over the hipbone and the outer surface of the bone itself are numbed with local anesthesia. Then, a special needle is inserted into the hipbone and about 1 tablespoon of bone marrow is drawn into a syringe. Another needle is inserted into the same area to collect a small piece of the bone marrow. Additional procedures may include allergen testing, urinalysis, and 24-hour urine collection.

Participants will return to NIH for reassessment of disease status in 12 to 18 months. The follow-up evaluation will include a history and physical examination, blood tests, possible repeat bone marrow and aspiration in patients whose clinical signs or symptoms change significantly, and other tests as clinically indicated.

First-degree relatives (parents, children, siblings) may be enrolled in limited instances to provide a blood sample for genetic analysis related to mast cell development and function for comparison with that of patients when they have similar symptoms.

DETAILED DESCRIPTION:
Anaphylaxis is a severe systemic hypersensitivity reaction caused by release of mediators from mast cells and basophils. Signs and symptoms of anaphylaxis may include generalized flushing, hives, stuffy nose, red and itchy eyes, difficulty in breathing, swelling of the tongue, throat, palms and soles, gastrointestinal cramping, lightheadedness and loss of consciousness. Although most common causes of anaphylaxis include foods, drugs and stinging insects, a causative factor is not identified in up to 50% of the patients with recurrent anaphylactic episodes. Mast cells are important mediators of anaphylaxis. This study will examine the hypothesis that some patients with unexplained anaphylaxis may have systemic mastocytosis, a disorder of pathologic mast cell proliferation, as an underlying cause. In addition, it will investigate hematopoietic cells, which result in their tissue mast cells being more susceptible to degranulation. The study will enroll patients with mastocytosis with or without flushing or anaphylaxis, and patients with unexplained flushing or anaphylaxis. Patients will receive a clinical evaluation, blood tests and a bone marrow biopsy and aspirate. Research studies planned include flow cytometric analysis of blood and bone marrow cells, investigation of mutations or polymorphisms in genes involved in mast cell growth and differentiation, determination of surrogate disease markers and examination of mast cell growth and function. The study will improve the understanding of the mechanisms involved in anaphylactic reactions, which could in turn lead to development of strategies to better prevent or treat the episodes.

ELIGIBILITY:
INCLUSION CRITERIA FOR PATIENTS WITH MASTOCYTOSIS:

Age equal to or greater than 18 years.

Diagnosis of mastocytosis established by presence of typical urticaria pigmentosa skin lesions or a bone marrow biopsy.

Letter of referral from prospective study participant's local doctor.

Ability to give informed consent.

EXCLUSION CRITERIA FOR PATIENTS WITH MASTOCYTOSIS:

Age less than 18 years.

Lack of a referral physician.

Presence of co-morbid conditions which, in the judgment of the investigator or the referring physician, may put the patient at undue risk for travel (such as an acute infection, severe thrombocytopenia).

Inability to provide informed consent.

Inability or refusal to undergo a bone marrow biopsy and aspirate.

Known allergy to latex or Lidocaine.

INCLUSION CRITERIA FOR PATIENTS WITH UNEXPLAINED FLUSHING OR ANAPHYLAXIS:

Age equal to or greater than 18 years.

Presence of flushing or anaphylaxis with negative workup for known causes such as carcinoid syndrome, pheochromocytoma, food allergy.

Ability to give informed consent.

EXCLUSION CRITERIA FOR PATIENTS WITH UNEXPLAINED FLUSHING OR ANAPHYLAXIS:

Same as for patients with mastocytosis.

Known cause for anaphylaxis or flushing.

Frequent life-threatening anaphylactic episodes: History of 6 or more separate attacks resulting in ER visits in the 6 months preceding the referral.

INCLUSION CRITERIA FOR RELATIVE:

To have a first-degree relative accepted to the protocol as a patient with unexplained anaphylaxis, flushing or mastocytosis.

Ability to give informed consent. For minors, ability of the parent to give informed consent.

There are no age restrictions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2002-10; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Neugut AI, Ghatak AT, Miller RL. Anaphylaxis in the United States: an investigation into its epidemiology. Arch Intern Med. 2001 Jan 8;161(1):15-21. doi: 10.1001/archinte.161.1.15. PMID 11146694
- [Background] Akin C, Kirshenbaum AS, Semere T, Worobec AS, Scott LM, Metcalfe DD. Analysis of the surface expression of c-kit and occurrence of the c-kit Asp816Val activating mutation in T cells, B cells, and myelomonocytic cells in patients with mastocytosis. Exp Hematol. 2000 Feb;28(2):140-7. doi: 10.1016/s0301-472x(99)00145-9. PMID 10706069
- [Background] Yavuz AS, Lipsky PE, Yavuz S, Metcalfe DD, Akin C. Evidence for the involvement of a hematopoietic progenitor cell in systemic mastocytosis from single-cell analysis of mutations in the c-kit gene. Blood. 2002 Jul 15;100(2):661-5. doi: 10.1182/blood-2002-01-0203. PMID 12091362